CLINICAL TRIAL: NCT05348538
Title: Feasibility Study of the Medication Review With Follow up Service for Patients With Polypharmacy in Swiss Community Pharmacies
Acronym: MaJ?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Pharmaceutical Society of the Vaud Canton ("SVPh: Société Vaudoise de pharmacie") (Unknown); Canton of Vaud ("État de Vaud") (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MaJ?-Unisanté-2022-v2
Record Dates: First submitted 2022-03-24; First posted 2022-04-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Chronic Disease
Keywords: Chronic disease; Prescription drugs
MeSH Terms: conditions — Chronic Disease | interventions — Medication Review

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medication review with follow up or MaJ? for the acronym in french (Experimental): All the pharmacists accepting to participate in the study will perform the intervention.
  Interventions: Other: Medication review with follow up or MaJ? for the acronym in french

INTERVENTIONS:
Other: Medication review with follow up or MaJ? for the acronym in french — MaJ? service will involve a pharmacist-patient face-to-face consultation with a 6-months interval during the study, it includes:
  1. Educational training: pharmacists will attend a half a day course. They will inform pharmacy technicians of their tasks. They will also have available an online version of the training about the service and data collection.
  2. Service provision: before the pharmacist-patient consultation (pharmacy technicians review the medication to identify the prescribed medication included in the treatment plan and to remove expired or medications non taken by the patient), during (pharmacist assess potential drug related problem) and after the consultation (to send a medication management plan to patients and doctors).
  3. Practice change facilitation to support pharmacists: pharmacists will be follow-up by the research team during the study (1st, 2nd, 3rd, 6th, 12th and 15th months of the study) to support them through the delivery of the service.
  Other Names: Medication review

SUMMARY:
In Switzerland, it is estimated that 20,000 people are hospitalized each year as a result of drug related problems (DRP). Community pharmacies (CP) are well positioned to identify and manage such DRPs in a timely manner. In Switzerland, no pharmacy service that focus on the management of DRPs is currently recognized and remunerated. A new service, medication review with follow up (MaJ? for the acronym in french), has been developed. It is focused on DRPs related to self-medication and medication management at home and it includes a systematic review of the patient's treatment.

Objective: To evaluate the impact of the MaJ? service for adults with polypharmacy in Swiss CP for the identification and management of DRPs.

A pre-post intervention study will be carried out in CPs in the canton of Vaud for 15 months. Volunteer pharmacists will include adults with a prescription for at least four chronic and systemic drugs since at least three months. Trained pharmacists will conduct structured consultations with a 6-months interval during the study to deliver the service. The primary outcome is the identification and management of DRPs. Secondary outcomes are patients' knowledge about their treatments, number of expired medications and description of pharmaceutical interventions.

The study has been approved and will be supported by Department of Health and Social Affairs in the canton of Vaud and the Cantonal Health Authorities. The Ethics Committee (CER-VD) concluded that the study does not fall under the Human Research Act. It will begin in spring 2022 in 19 to 35 pharmacies that will recruit at least 162 patients after randomization of eligible patients through a sequence of computer-generated random numbers. Ad-hoc tools (medication management plan) and validated tools (PharmDISC tool, patient knowledge tool) will guide pharmacists throughout the consultation. Educational training and support for pharmacists will increase quality of service provision and fidelity of study protocol. A sub analysis will be carried out for those patients included who are 65 years old or over in order to target the intervention to a specific group of patients with higher risk for DRPs.

This study will evaluate the impact of a new service that includes validated, structured and standardized interventions, training and supervision for CP staff, non-prescription medication evaluation and use of home-based patient records. MaJ? is an enhanced service designed to overcome those barriers found in the implementation process of medication review services.

DETAILED DESCRIPTION:
1. Background

   1.1. Role of the pharmacist: The role of the community pharmacist includes an increasing number of responsibilities. Whereas in the past the aspects related to the manufacture and sale of medicines were predominant, the 2000s saw the emergence of other roles for the pharmacist in Switzerland, primarily in order to control rising health care costs. With the implementation of the remuneration based on services (RBP for the french acronym) in 2001, a step forward was taken in the direction of pharmaceutical services, for example by the remuneration of the pharmaceutical record during the delivery of prescribed medicines. Since 2001, the RBP has been amended several times in order to respond to the health care system needs and the activities of community pharmacists in relation to patients' needs (adherence, poly-medication, etc.).

   According to the Federal Council, pharmacists could still take on additional tasks in the field of primary care, as they offer easier access to health advice. Since 2016, the "Grand Conseil du Canton de Vaud" has been supporting the implementation of a shared medication plan concerning "medication safety throughout the care process". The aim is to evaluate the implementation of a collaborative management of patients' treatment based on the e-health platform for the canton of Vaud on poly-medicated patients with multiple carers (general medical practitioners -GP-, community pharmacies -CP- and nursing homes). In this context, new opportunities exist to strengthen the role of the pharmacist in the care process. In addition to prescribed medications, pharmacists also advise patients when they self-medicate. Self-medication is "the selection and use of medication, including herbal and traditional products, by individuals to treat symptoms or diseases that they have identified themselves". Community pharmacists are often the first health professionals to be contacted by patients with minor ailments. In order to ensure responsible self-medication with non-prescription medication, pharmacist advice is necessary.

   Therefore, community pharmacists are in a privileged position to have an overview of all the medicines taken by patients (prescription and non-prescription). A study carried out in the Canton of Vaud in 2017 with diabetic patients showed that 79% of them had visited only one pharmacy in the last 12 months (96% two pharmacies maximum).

   1.2. Drug-related problems (DRPs): The Pharmaceutical Care Network Europe (PCNE) describes a DRP as "an event or circumstance involving drug therapy that actually or potentially interferes with the expected optimal outcome of medical care". The PCNE has developed a classification of DRPs that has evolved over time and among investigators. Thus, the variation in classifications makes it difficult to standardize this topic, especially on a more accurate description of the clinical and economic burden of DRP.

   As an example, it has been estimated that the costs of DRP such as non-adherence is approximately 125 billion euro per year in the European Union. In Switzerland, each year, 20,000 hospitalizations result from DRP. DRPs have several causes, whether related to the patient or to the health process. For example, if the patient is not familiar with his/her treatment, he/she will not be motivated to take it, especially if the disease is chronic and the symptoms are not obvious. In this situation, an adherence problem could arise resulting in health care costs (hospitalizations, medical visits, etc.) that could have been avoided.

   Another example of DRP could be a treatment intake error (inadequate posology, etc.) due to a drug package that is misunderstood or missing or due to old medication storage at home. Intake errors could lead to a decrease of treatment effectiveness or to an increase in adverse effects and risks of drug interactions.

   Another example of DRP could be inadequate storage of medicaments. Treatments such as eye drops could lead to eye infections if they are not properly storage. Similarly, improperly stored insulin pens could lose their effectiveness due to a decrease in insulin concentration.

   These sources of DRP can be prevented and managed through pharmaceutical interventions. A pharmaceutical intervention is described as "any action performed by the pharmacist that result in a change in treatment or therapy management". It is well known that pharmaceutical interventions, such as patient counseling, can reduce DRP.

   One way to identify and prevent the occurrence of DRP in a structured manner is to conduct a medication review with the patient.

   To document community pharmacists' clinical activities, including the identification and management of DRPs, a tool was developed and validated in Swiss CPs.

   1.3. Medication Review: Medication review is defined as "a structured evaluation of the patient's medications with the goal of optimizing their use and improving health status", it involves the detection of DRPs and the recommendation of interventions.

   In Switzerland nowadays, the Swiss law details what pharmacists have to do in order to identify and manage DRPs at the time of the delivery of prescription medications to the patient (check for interactions, contraindications, dosage, etc.). However, there is no service that specifically targets the identification and management of DRPs possibly induced by the patients (adherence, wrong conservation, missing or forgotten information, etc.). The Cantonal Health Authorities set up the project (medication review with follow up or MaJ? for the acronym in french) in collaboration with the Center for Primary Care and Public Health of the University of Lausanne (Unisanté) and the Department of Health and Social Affairs in the canton of Vaud. The aim of the MaJ? service is to perform a medication review at the CP to: 1) achieve a decrease in the number of DRPs, 2) improve patients' literacy about their treatments and 3) remove of expired medications for proper elimination by the CPs. This service allows the pharmacists going further than usual prescription validation in terms of detection of DRPs and pharmaceutical interventions. Based on the principles of the "brown bag" (medication review first described in 1982 in the United States) and medication review with follow up, MaJ? includes all the treatments consumed by the patient (prescribed and non-prescribed medication), who brings them to the CP before performing the service. MaJ? is a service that offers several advantages: first, the material aims to guide and facilitate the detection of DRPs through the use of a validated tool and to record pharmaceutical interventions as well as offering information to the prescribing GP. This service also offers patients a review of self-medication (non-prescription medication). MaJ? strengthens the role of pharmacy technicians to perform an initial sorting of the medication brought to the CP to eliminate expired drugs, to allow the pharmacist an optimal use of the time devoted to the consultation. The service is in line with the national objective to reinforce pharmacy technicians' role, their education and to allow them to assist (under supervision) some services.

   1.4. PharmDISC tool: PharmDISC is a standardised classification system of DRPs and pharmaceutical interventions. The tool was validated in 2014 in Swiss CPs (PI) and it was based on a existing hospital system (the Swiss Association of Public Health Administration and Hospital Pharmacists - GSASA). Community pharmacist who tested the system agreed that "documentation should enhance traceability and information flow within team and with other healthcare professionals, improving so the visibility of pharmacists' activities".
2. Objectives The purpose of the study is to evaluate the feasibility and impact of the MaJ? service for adults with polypharmacy in CP in the canton of Vaud (Switzerland).

   Primary objectives To evaluate the impact of MaJ? on the identification and management of DRP. Secondary objectives To assess the impact of MaJ? on the number of expired medications. To assess the impact of MaJ? on patients' knowledge about their treatments. To describe the interventions made by the pharmacists through MaJ?.
3. Method

   3.1. Research design Pre-post intervention study carried out in Swiss CPs from the canton of Vaud. Each CP will be considered a cluster to avoid contamination. The study will take place over 15 months between spring 2022 and summer 2023.

   3.2. Participants enrollment

   3.2.1. Pharmacies and pharmacists The Cantonal Health Authorities and the Department of Health and Social Affairs in the canton of Vaud will provide CPs with the study information via email.

   In order to participate in this study, pharmacies must meet the following criteria:
   * Employ at least one pharmacist who has completed the MaJ? training to perform the service.
   * Name a pharmacist as the contact pharmacist, who agrees to represent the pharmacy for communication purposes with the research team and for submitting study data.
   * To include at least one patient in the study.

   In order to participate in this study, pharmacists must meet the following criteria:
   * Participate in MaJ? training session.
   * Give oral consent to participate in the research study. The same community pharmacist may care for multiple patients but each patient has to be taken care of by the same-trained pharmacist at each consultation. A pharmacist who works in different participating pharmacies will be assigned to the pharmacy where he/she works higher number of hours per week. After initial training, new eligible pharmacists who start working in participant pharmacies will be able to participate if complete the online training.

   Pharmacists will receive a remuneration of 100 Swiss Francs per review (which cannot be financed by the basic health insurance) for the additional time spent on the research during each documented consultation according to the guidelines in the educational training.

   During patient enrollment, pharmacists will be contacted by the research team to keep them informed of recruitment progress and to motivate them to enroll new patients. These contacts will be made by phone and email.

   3.2.2. Patients: inclusion criteria for patients are included below. The CP will send the list of patients in the CP with the inclusion criteria (this list will not include patients' identification but CP codes). In order to avoid selection bias during recruitment, a member of the research team will randomize 50 patients from the list (randomized through a sequence of computer-generated random numbers). The research team will send an inclusion form to the contact pharmacist of each CP with the 50 patients randomized for them to contact the patients by phone or in person in CP and fill it with the information provided by patients. Participating pharmacists will be asked to enroll at least one to ten patients.

   3.2.3. Sample size calculation Primary objective of the study aims to measure the difference in DRPs per patient observed between the first and second consultation with the patient, and the first and third consultation with the patient. Sample size calculation was based on this primary study outcome to detect a difference of 0.5 DRPs per patient at the end of the study. The sample size was calculated with ≥0.8 power, type I error rate of 5%, assuming an intra-cluster correlation of 0.02. Allowing for 15% dropout, the overall sample size is 162 patients, with 19 to 35 pharmacies (1-10 patients per CP).

   3.3. Description of the intervention

   3.3.1. Pharmacy staff training: Pharmacists will attend a half a day course (four hours) that will cover service provision, good practice standards, patients' recruitment, communication skills with patients and other health professionals, data collection and study protocol. The workshop will include a combination of lecture presentations and interactive sessions including role-play scenarios. The training will be evaluated and accredited for pharmacists' continuing professional development. Pharmacists will inform and train pharmacist's technicians for their tasks. They will also have available an online version of the training about the service and data collection.

   3.3.2. Practice change facilitator: Participant pharmacists will be follow-up by the research team via telephone during the study at least six times (1st, 2nd, 3rd, 6th, 12th and 15th months of the study) to support them through the delivery of the service. Pharmacists will also be able of contacting the research team by email throughout the study concerning service provision, data entry, etc. The facilitation process will be explained to pharmacists during the training session. Facilitation process allows ensuring recruitment targets are met, quality of service provision and fidelity to study protocol.

   3.3.3. Medication review with follow up

   Aims of the service: The aim of the service is to perform a medication review at the CP to achieve the following goals:
   * To remove expired medications.
   * To improve patients' knowledge about their treatments.
   * To decrease the number of DRPs.

   An intervention plan (sent to the GP) is developed based on the pharmacy record, treatments reported by the patient and the consultation. Patients are asked to bring all their medication to the pharmacy, where they are sorted by the pharmacy technician. The medication management plan is then reviewed and explained to the patient by the pharmacist. The pharmacist also checks to identify potential DRPs such as adherence issues and propose interventions to solve them.

   Then, the service is provided in three stages:

   Before the pharmacist-patient consultation. During the pharmacist-patient consultation at the CP. After the pharmacist-patient consultation at the pharmacy. The different tasks performed by the pharmacist or pharmacy technician are also differentiated.

   Procedure of MaJ?:

   - Before the pharmacist-patient consultation

   The purpose of this step is to prepare the necessary documents for the service before the appointment with the patient. The pharmacy technician pre-fills the documents with the following information:

   - Medication management plan: Patient data: for patient identification purposes by the pharmacy. Patient Id: pharmacy software codes. Pharmacy stamp. Medication data: treatment and prescriber information (name of drug prescribed, dose, posology and prescriber's name).

   - Removed medication form: Patient data: for patient identification purposes by the pharmacy. Patients' acceptance of the consultation. Eligibility to receive the benefit: determined by being adult, having four or more medications and the patient's agreement, which determines reimbursement. At the moment of the recruitment, eligible patients should still have inclusion criteria at the time of the first pharmacist-patient consultation. If, after the first pharmacist-patient consultation, a patient have any treatment change and inclusion criteria is no longer met, he/she can still be included in the service.

   Potential treatments to be removed: brand name/INN (international non-proprietary names), dose, formulation.

   Time: time spent by the pharmacy technician to prepare the documents. Medication by group: an initial medication review by the pharmacy technician is carried out. This can be accomplished by the patient bringing their own medications prior to the consultation or throughout other arrangements with the CP. The technician separates the patient's medications into two groups: Group I (prescribed-medication that are part of the medication plan), Group II (medication outside the medication plan, this could be over-the-counter drugs or medication not currently prescribed).

   Before patient's arrival, the pharmacist must have at least 30 minutes to review the patient's medications. The purpose of this review is to have the opportunity to assess potential DRPs and to list them using the PharmDISC tool.

   During the pharmacist-patient consultation The purpose of this consultation is to discuss the potential DRPs and to evaluate and improve patient's knowledge of his/her treatment using the patient's medication knowledge evaluation tool. The pharmacist proposes different interventions to the patient to resolve identified DRPs. This is done using the PharmDISC tool. Patient's non-prescription medications are briefly discussed during this encounter to resolve patients' questions. The pharmacist gives advice about the disposal of expired or unused medications. Pharmacists can also add comments to each page of the forms.

   Pharmacists and patients should sign the forms for compensation purposes. After the pharmacist-patient consultation: The purpose of this phase is to inform the GP by providing report of the consultation with the patient and the medication management plan. In case of different GPs prescribing treatments to the patient, this report may improve communication between health care practitioners and patient's management.

   After the consultation, within a maximum of two-day' period, the pharmacist completes the medication management plan, with medicaments from groups I and II, according to that discussed with the patient. If a pharmacy already has a standard practice form, the pharmacist can use it while following instructions given.

   The medication management plan is given to both, patient and GP. However, in case of discrepancies between the medication record and the medication brought in by the patient, the pharmacist can forward the form to the GP for validation before handing it to the patient. In addition, the pharmacist should complete a medication review report, describing the identified DRPs relevant to the GP and the interventions taken to manage and/or resolve them. This report is also sent to the GP. The report should also be sent to the GP within a maximum of two-day' period after the pharmacist-patient consultation.

   Time frame for the intervention: Pharmacists must carry out three different consultations with the patients with a 6-months interval, at the beginning, six months later and 12 months after the first encounter. The first pharmacist-patient consultation will take place after patient recruitment. After anonymizing data, contact pharmacists in each pharmacy will send a copy of the information to the research team (within one month after the first consultation) The second pharmacist-patient consultation will take place 6 months after the first consultation. The intervention will be conducted similarly to the first consultation and using the same forms. Copy of data will be provided to the research team within one month after completing the second consultation. The third pharmacist-patient consultation will take place 12 months after the first one. The intervention will be conducted similarly to the first and second consultation and using the same forms. Copy of data will be provided to the research team within one month after completing the last consultation.

   3.4. Data analysis Continuous variables will be reported using mean and standard deviation, or median and percentiles depending on the distribution of the variable (the Kolmogorov Smirnov test will be used to assess normality). Categorical variables will be reported using frequency and proportion. For the comparison of continuous variables, the T Student's test or the ANOVA test will be carried out if there is a normal distribution, and Kruskal-Wallis otherwise. The comparison of the categorical variables will be carried out using the χ2 test, the Fisher's exact test or Yate's chi-squared test if necessary.

   For each patient under study, differences between consultations will be compared for dependent variables (DRPs, pharmaceutical interventions, pharmaceutical interventions acceptance, patient knowledge, medication removed). A linear regression model will be performed accounting for the cluster effect. Firstly, variables will be considered significant (p-value<0.2) in a bivariate model to be included in a multivariate model. Secondly, the variables considered significant at a value of p<0.1 in the multivariate model will be included in the final model. The level of significance will be set at p<0.05, the software STATA® will be used.

   An analysis with completed cases will be made. In addition, an analysis with the whole sample will be made where, for the management of missing data, initial value will be considered as not been modified (baseline observation carried forward-BOCF). A sub analysis will be carried out for those patients included who are 65 years old or over in order to target the intervention to a specific group of patients with higher risk for DRPs.

   3.5. Data handling Participating pharmacists are responsible for keeping all documents in the CP according to current practices and requirements.

   Different forms used during the study will be collected in paper or electronic format (e-mail) through the contact pharmacists. Research team at Unisanté will code data in a database specifically designed for the study. Data will only be accessible by researchers involved in the project and will be hosted on Unisanté's server (backed up electronically). At the end of the study, data will be kept up to 10 years after the last publication.
4. Data confidentiality and ethical aspects According to the Cantonal Commission for Ethics in Human Research (CER-VD), this study does not fall under the Human Research Act (HRA), therefore, this protocol does not need to be submitted for review. Participants will not need to sign a consent form. Patients' signatures will be requested as proof of service provision and, if necessary, for transmission of the medication plan to the GP.

   The information will be coded, anonymized and the data will be referenced by assigned numbers for both the published and non-published information. All the information collected will be stored in the repository of Unisanté, being accessible only to authorized personnel.
5. Medical monitoring and insurance The service is considered to fall under usual practice of CP, the aim of the service proposed is to give structure to this usual practice, therefore there is no need for safety considerations nor additional insurance. Pharmacists will be able to continue to provide routine care to patients about DRP management. Therefore, no special medical supervision is required. Pharmacists are free to contact GPs in agreement with patients as usual.
6. Financial support Public-private partnership Cantonal Health Authorities - Department of Health and Social Affairs in the canton of Vaud provides for a reimbursement of 100 Swiss Francs per pharmacist-patient consultation. There is no compensation for patients included.
7. Conflict of interest No conflicts of interest are declared. However, the investigators are committed to the development of services within their professional competencies. They are committed to handle data in a rigorous and transparent manner to avoid bias in the collecting, interpretation and discussion of the results.
8. Dissemination plan The findings obtained after the study will be disseminated through the usual methods of scientific dissemination, including communications to congresses and publications in scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a prescription for at least four chronic and systemic drugs for at least the last three months.

Exclusion Criteria:

* Patients suffering from dementia, psychiatric disorder, or other health condition that hinders obtaining informed consent and/or conducting the consultations with the pharmacist.
* Patients who disagree meeting the pharmacist for the three consultations during the study with a 6-months interval.
* Patients who are not able to bring all their medication to the community pharmacy.
* Patients who cannot speak and read French.
* Patients who does not allow the pharmacist contacting the general medical practitioner to inform him/her about possible drug related problems.
* Patients who will not consent of participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in number of drug related problems (DRPs) | At three points during the study: 1. First pharmacist-patient consultation, 2. Second consultation (6 months after the first one) and 3. Third consultation (12 months after the first one).
  Number of DRPs detected by the pharmacist during the pharmacist-patient consultation. Pharmacists will complete the management plan and PharmDISC tool at all consultations with the patient (three consultations with a 6-months interval). It will be assessed by comparing the differences between the first and second consultations and the first and third consultations. Total number of DRP and mean per patient will be calculated.
Change in DRPs | At three points during the study: 1. First pharmacist-patient consultation, 2. Second pharmacist-patient consultation (6 months after the first one) and 3. Third pharmacist-patient consultation (12 months after the first one)
  Pharmacists will complete the PharmDISC tool which includes:
  1. Therapy choice: no concordance with guidelines, contraindication, interaction, drug not indicated, duplication, adverse effect, incomplete patient documentation.
  2. Drug choice: inappropriate dosage form.
  3. Dose choice: underdose/overdose, inappropriate monitoring, dose not adjusted to organ function.
  4. Drug use: inappropriate timing of frequency of administration, inappropriate use method.
  5. Therapy duration: inappropriate therapy duration.
  6. Logistics: prescribed drug not available, error in medication process.
  7. Patient: insufficient adherence, insufficient knowledge, burden due to therapy.
  8. Other PharmDISC tool has also classification related to health problems: treatment effectiveness, untreated indication, safety of treatment, treatment costs, dissatisfaction/problems of the patient.
  PharmDISC tool has also classification related to type of problem: manifest, potential.

SECONDARY OUTCOMES:
Change in number of medications removed | At three points during the study: 1. First pharmacist-patient consultation, 2. Second pharmacist-patient consultation (6 months after the first one) and 3. Third pharmacist-patient consultation (12 months after the first one)
  Medication expired or non taken by the patient. This can be accomplished after reviewing the medication brought by the patient to the pharmacy. Total number, mean per patient and percentage in relation to the total medication brought by the patient and accepted by the patient to be removed after pharmacist-patient consultation.
Change in patients' knowledge | At three points during the study: 1. First pharmacist-patient consultation, 2. Second pharmacist-patient consultation (6 months after the first one) and 3. Third pharmacist-patient consultation (12 months after the first one)
  Medication knowledge evaluation tool with 4 questions (medication cited/medication known/why taking the medication/posology known). The patient scores 1 point if he/she knows the correct answer and 0 points if he/she does not know. Score goes from 0 (patient does not know the medication) to 4 (patient completely knows the medication) for each medication that the patient is taking.
Change in number of pharmaceutical interventions | At three points during the study: 1. First pharmacist-patient consultation, 2. Second pharmacist-patient consultation (6 months after the first one) and 3. Third pharmacist-patient consultation (12 months after the first one)
  Number of interventions carried out by the pharmacist with patients and/or general medical practitioners to solve drug related problems.
Change in pharmaceutical interventions | At three points during the study: 1. First pharmacist-patient consultation, 2. Second pharmacist-patient consultation (6 months after the first one) and 3. Third pharmacist-patient consultation (12 months after the first one)
  Classification of interventions will be made by the pharmacist using the PharmDISC tool:
  * Counselling of patient
  * Application instruction (training)
  * Delivery of an adherence aid (ex. pill box) inclusive counselling
  * Therapy started
  * Therapy stopped/no delivery
  * Substitution
  * Dose adjustment
  * Therapy monitoring
  * Optimization of administration
  * Change of administration way
  * Adjustment of the delivery amount (package size, quantity of packages, etc.)
  * Information to the GP
  * Clarification in the case notes (history)
  * Report to pharmacovigilance center
  * Other

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Berger, PhD, Study Chair — Unisanté
Locations (1):
- Unisanté, Center of Primay Care and Public Health, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Septembre 2023 - August 2024
Access Criteria: Contact principal investigator.

REFERENCES:
- [Background] Guignard E, Bugnon O. Pharmaceutical care in community pharmacies: practice and research in Switzerland. Ann Pharmacother. 2006 Mar;40(3):512-7. doi: 10.1345/aph.1G199. Epub 2006 Feb 7. PMID 16467249
- [Background] Hersberger KE, Messerli M. Development of Clinical Pharmacy in Switzerland: Involvement of Community Pharmacists in Care for Older Patients. Drugs Aging. 2016 Mar;33(3):205-11. doi: 10.1007/s40266-016-0353-6. PMID 26884391
- [Background] Krahenbuhl JM, Kremer B, Guignard B, Bugnon O. Practical evaluation of the drug-related problem management process in Swiss community pharmacies. Pharm World Sci. 2008 Dec;30(6):777-86. doi: 10.1007/s11096-008-9217-4. Epub 2008 Apr 6. PMID 18392732
- [Background] Lim XY, Yeo QQ, Kng GLL, Chung WL, Yap KZ. Validation of a Drug-Related Problem Classification System for the Intermediate and Long-Term Care Setting in Singapore. Pharmacy (Basel). 2018 Oct 3;6(4):109. doi: 10.3390/pharmacy6040109. PMID 30282930
- [Background] Vrijens B, Antoniou S, Burnier M, de la Sierra A, Volpe M. Current Situation of Medication Adherence in Hypertension. Front Pharmacol. 2017 Mar 1;8:100. doi: 10.3389/fphar.2017.00100. eCollection 2017. PMID 28298894
- [Background] Perez-Jover V, Mira JJ, Carratala-Munuera C, Gil-Guillen VF, Basora J, Lopez-Pineda A, Orozco-Beltran D. Inappropriate Use of Medication by Elderly, Polymedicated, or Multipathological Patients with Chronic Diseases. Int J Environ Res Public Health. 2018 Feb 10;15(2):310. doi: 10.3390/ijerph15020310. PMID 29439425
- [Background] Dooley MJ, Allen KM, Doecke CJ, Galbraith KJ, Taylor GR, Bright J, Carey DL. A prospective multicentre study of pharmacist initiated changes to drug therapy and patient management in acute care government funded hospitals. Br J Clin Pharmacol. 2004 Apr;57(4):513-21. doi: 10.1046/j.1365-2125.2003.02029.x. PMID 15025751
- [Background] Hanlon JT, Lindblad CI, Gray SL. Can clinical pharmacy services have a positive impact on drug-related problems and health outcomes in community-based older adults? Am J Geriatr Pharmacother. 2004 Mar;2(1):3-13. doi: 10.1016/s1543-5946(04)90002-5. PMID 15555474
- [Background] Tasaka Y, Tanaka A, Yasunaga D, Asakawa T, Araki H, Tanaka M. Potential drug-related problems detected by routine pharmaceutical interventions: safety and economic contributions made by hospital pharmacists in Japan. J Pharm Health Care Sci. 2018 Dec 13;4:33. doi: 10.1186/s40780-018-0125-z. eCollection 2018. PMID 30564432
- [Background] Messerli M, Blozik E, Vriends N, Hersberger KE. Impact of a community pharmacist-led medication review on medicines use in patients on polypharmacy--a prospective randomised controlled trial. BMC Health Serv Res. 2016 Apr 23;16:145. doi: 10.1186/s12913-016-1384-8. PMID 27108410
- [Background] Griese-Mammen N, Hersberger KE, Messerli M, Leikola S, Horvat N, van Mil JWF, Kos M. PCNE definition of medication review: reaching agreement. Int J Clin Pharm. 2018 Oct;40(5):1199-1208. doi: 10.1007/s11096-018-0696-7. Epub 2018 Aug 2. PMID 30073611
- [Background] Messerli M, Vriends N, Hersberger KE. Humanistic outcomes and patient acceptance of the pharmacist-led medication review "Polymedication Check" in primary care in Switzerland: a prospective randomized controlled trial. Patient Prefer Adherence. 2018 Jun 19;12:1071-1078. doi: 10.2147/PPA.S160789. eCollection 2018. PMID 29950820
- [Background] Rutter P. Role of community pharmacists in patients' self-care and self-medication. Integr Pharm Res Pract. 2015 Jun 24;4:57-65. doi: 10.2147/IPRP.S70403. eCollection 2015. PMID 29354520
- [Background] Cooper RJ. Over-the-counter medicine abuse - a review of the literature. J Subst Use. 2013 Apr;18(2):82-107. doi: 10.3109/14659891.2011.615002. Epub 2011 Oct 3. PMID 23525509
- [Background] Maes KA, Hersberger KE, Lampert ML. Pharmaceutical interventions on prescribed medicines in community pharmacies: focus on patient-reported problems. Int J Clin Pharm. 2018 Apr;40(2):335-340. doi: 10.1007/s11096-018-0595-y. Epub 2018 Feb 5. PMID 29404780
- [Background] Nathan A, Goodyer L, Lovejoy A, Rashid A. 'Brown bag' medication reviews as a means of optimizing patients' use of medication and of identifying potential clinical problems. Fam Pract. 1999 Jun;16(3):278-82. doi: 10.1093/fampra/16.3.278. PMID 10439982
- [Background] O'Connell MB, Chang F, Tocco A, Mills ME, Hwang JM, Garwood CL, Khreizat HS, Gupta NS. Drug-Related-Problem Outcomes and Program Satisfaction from a Comprehensive Brown Bag Medication Review. J Am Geriatr Soc. 2015 Sep;63(9):1900-5. doi: 10.1111/jgs.13597. Epub 2015 Aug 27. PMID 26313706
- [Background] Sarzynski EM, Luz CC, Rios-Bedoya CF, Zhou S. Considerations for using the 'brown bag' strategy to reconcile medications during routine outpatient office visits. Qual Prim Care. 2014;22(4):177-87. PMID 25695529
- [Background] Ocampo CC, Garcia-Cardenas V, Martinez-Martinez F, Benrimoj SI, Amariles P, Gastelurrutia MA. Implementation of medication review with follow-up in a Spanish community pharmacy and its achieved outcomes. Int J Clin Pharm. 2015 Oct;37(5):931-40. doi: 10.1007/s11096-015-0145-9. Epub 2015 Jun 4. PMID 26040837
- [Background] Varas-Doval R, Gastelurrutia MA, Benrimoj SI, Garcia-Cardenas V, Saez-Benito L, Martinez-Martinez F. Clinical impact of a pharmacist-led medication review with follow up for aged polypharmacy patients: A cluster randomized controlled trial. Pharm Pract (Granada). 2020 Oct-Dec;18(4):2133. doi: 10.18549/PharmPract.2020.4.2133. Epub 2020 Oct 21. PMID 33149794
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] de Barra M, Scott C, Johnston M, De Bruin M, Scott N, Matheson C, Bond C, Watson M. Do pharmacy intervention reports adequately describe their interventions? A template for intervention description and replication analysis of reports included in a systematic review. BMJ Open. 2019 Dec 19;9(12):e025511. doi: 10.1136/bmjopen-2018-025511. PMID 31862736
- [Background] McPherson ML, Smith SW, Powers A, Zuckerman IH. Association between diabetes patients' knowledge about medications and their blood glucose control. Res Social Adm Pharm. 2008 Mar;4(1):37-45. doi: 10.1016/j.sapharm.2007.01.002. PMID 18342821
- [Background] Liu-Seifert H, Zhang S, D'Souza D, Skljarevski V. A closer look at the baseline-observation-carried-forward (BOCF). Patient Prefer Adherence. 2010 Feb 4;4:11-6. doi: 10.2147/ppa.s8135. PMID 20165594
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Okuyan B, Sancar M, Izzettin FV. Assessment of medication knowledge and adherence among patients under oral chronic medication treatment in community pharmacy settings. Pharmacoepidemiol Drug Saf. 2013 Feb;22(2):209-14. doi: 10.1002/pds.3275. Epub 2012 Apr 18. PMID 22514147
- [Background] Jokanovic N, Tan EC, Sudhakaran S, Kirkpatrick CM, Dooley MJ, Ryan-Atwood TE, Bell JS. Pharmacist-led medication review in community settings: An overview of systematic reviews. Res Social Adm Pharm. 2017 Jul-Aug;13(4):661-685. doi: 10.1016/j.sapharm.2016.08.005. Epub 2016 Aug 28. PMID 27665364
- [Background] Malet-Larrea A, Goyenechea E, Garcia-Cardenas V, Calvo B, Arteche JM, Aranegui P, Zubeldia JJ, Gastelurrutia MA, Martinez-Martinez F, Benrimoj SI. The impact of a medication review with follow-up service on hospital admissions in aged polypharmacy patients. Br J Clin Pharmacol. 2016 Sep;82(3):831-8. doi: 10.1111/bcp.13012. Epub 2016 Jun 9. PMID 27195696
- [Background] Varas-Doval R, Gastelurrutia MA, Benrimoj SI, Zarzuelo MJ, Garcia-Cardenas V, Perez-Escamilla B, Martinez-Martinez F. Evaluating an implementation programme for medication review with follow-up in community pharmacy using a hybrid effectiveness study design: translating evidence into practice. BMJ Open. 2020 Sep 29;10(9):e036669. doi: 10.1136/bmjopen-2019-036669. PMID 32994235
- [Background] Noain A, Garcia-Cardenas V, Gastelurrutia MA, Malet-Larrea A, Martinez-Martinez F, Sabater-Hernandez D, Benrimoj SI. Cost analysis for the implementation of a medication review with follow-up service in Spain. Int J Clin Pharm. 2017 Aug;39(4):750-758. doi: 10.1007/s11096-017-0454-2. Epub 2017 Apr 22. PMID 28434119
- [Background] Jodar-Sanchez F, Malet-Larrea A, Martin JJ, Garcia-Mochon L, Lopez Del Amo MP, Martinez-Martinez F, Gastelurrutia-Garralda MA, Garcia-Cardenas V, Sabater-Hernandez D, Saez-Benito L, Benrimoj SI. Cost-utility analysis of a medication review with follow-up service for older adults with polypharmacy in community pharmacies in Spain: the conSIGUE program. Pharmacoeconomics. 2015 Jun;33(6):599-610. doi: 10.1007/s40273-015-0270-2. PMID 25774017
- [Background] Ahumada-Canale A, Vargas C, Martinez-Mardones F, Plaza-Plaza JC, Benrimoj S, Garcia-Cardenas V. Cost-utility analysis of medication review with follow-up for cardiovascular outcomes: A microsimulation model. Health Policy. 2021 Nov;125(11):1406-1414. doi: 10.1016/j.healthpol.2021.09.004. Epub 2021 Sep 16. PMID 34579954
- [Background] Stratton SJ. Quasi-Experimental Design (Pre-Test and Post-Test Studies) in Prehospital and Disaster Research. Prehosp Disaster Med. 2019 Dec;34(6):573-574. doi: 10.1017/S1049023X19005053. No abstract available. PMID 31767051
- [Derived] Amador-Fernandez N, Escaith M, Simi E, Quintana-Barcena P, Berger J. Evaluation of an enhanced service for medication review with follow up in Swiss community pharmacies: Pre-post study protocol. PLoS One. 2023 Oct 17;18(10):e0292037. doi: 10.1371/journal.pone.0292037. eCollection 2023. PMID 37847695
- See also: Vaud Éd. Exposé des motifs et projet de décret sur le développement d'outils et de processus favorisant la continuité et la coordination des soins. Canton de Vaud: État de Vaud 2016 — https://www.vd.ch/toutes-les-autorites/grand-conseil/seances-precedentes/annee-2016/seance-du-mardi-6-et-mercredi-7-decembre-2016/expose-des-motifs-et-projet-de-decret-sur-le-developpement-doutils-et-de-processus-favorisant-la-continuite-et-la-coordination-des-soins/.
- See also: Fedlex. RS 811.11 Loi fédérale du 23 juin 2006 sur les professions médicales universitaires: Confédération Suisse. ; 2021 — https://www.admin.ch/opc/fr/classified-compilation/20040265/index.html.
- See also: NICE. Medicines optimisation: the safe and effective use of medicines to enable the best possible outcomes. www.nice.org.uk/guidance/ng5: Nice Institute for Health and Care Excellence; 2015 — https://www.nice.org.uk/guidance/ng5
- See also: FIP. Empowering self-care: A handbook for pharmacists. . The Hague: International Pharmaceutical Federation 2022. — https://www.fip.org/file/5111
- See also: WHO. Classification of self-care interventions for health: a shared language to describe the uses of self-care interventions. Geneva: World Health Organization; 2021. — https://www.who.int/publications/i/item/9789240039469